CLINICAL TRIAL: NCT04716049
Title: The Effectiveness of Two Different Combinations of Recovery Methods in Elite Professional Young Soccer Players: a RCT
Brief Title: Effectiveness of Recovery Protocols in Elite Professional Young Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RCTREC001
Record Dates: First submitted 2021-01-12; First posted 2021-01-20 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Soccer; Physical Stress; Fatigue
Keywords: performance; recovery; fatigue; soccer
MeSH Terms: conditions — Fatigue | interventions — somatostatin, cyclic hexapeptide(Phe-Phe-Trp-Lys-Thr-Phe)-

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol I (Experimental): Powerade© Carbohydrates+Protein Cherry Juice Foam Roller Cold Water Immersion
  Interventions: Other: Powerade©, CHP, CJ, FR, CWI
- Protocol II (Experimental): Powerade@ Carbohydrates+Protein Stretching Intermittent Cold-Water Immersion
  Interventions: Other: Powerade©, CHP, STR, ICWI

INTERVENTIONS:
Other: Powerade©, CHP, CJ, FR, CWI — Combination of recovery strategies including dietary, neuromuscular and physiological as follows:
  Powerade©: players will drink 500 mL during the game
  Carbohydrate and protein (CHP): players will drink 250 mL of water with CHP within 30 minutes after the end of the game.
  Tart cherry concentrate (CJ): players will drink 30 mL of CJ within 30 minutes after the end of the game.
  Foam roller (FR): players will follow FR protocol using a polyvinylchloride pipe roller. They will begin with the FR at the most proximal portion of the muscle and to roll as much body mass as tolerable back and forth at a cadence of 1 second superior and 1 second inferior for 45 seconds followed by a 15-second rest for each muscle group (quadriceps, adductors, hamstrings, abductors and calf) in each extremity and repeated once.
  Cold Water Immersion (CWI): will be the last strategy used. Players will immerse their lower body to the level of hips for 10 minutes in cold water (13-14°C).
  Arms: Protocol I
Other: Powerade©, CHP, STR, ICWI — Combination of recovery strategies including dietary, neuromuscular and physiological as follows:
  Powerade©: players will drink 500 mL of "Powerade©" during the game
  Carbohydrate and protein intake (CHP): players will drink 250 mL of water with CHP within 30 minutes after the end of the competition.
  Stretching (STR): players will perform 10-min of static stretching, involving 2 unilateral repetitions of 30 seconds held stretches to the quadriceps, adductors, hamstrings, abductors and calf muscles.
  Intermittent Cold-Water Immersion (ICWI): will be the last strategy used. It will consist of five 2 min intermittent immersions of the lower limb (up to the iliac crest) in a cold-water bath (13-14ºC), separated by 2 min rest in ambient air. Ice will be added to the bath at regular intervals to maintain water temperature at 13-14ºC. Players will be instructed to stand in the bath, with as little movement as possible.
  Arms: Protocol II

SUMMARY:
The main objective of this project is to compare two recovery protocols, including nutritional and neuromuscular strategies on inmune, physiological and muscular responses.

DETAILED DESCRIPTION:
A randomized controlled trial will be performed and players will be assigned in one of the two groups after their participation in a football game. The investigators will take baseline measures before the game and post-competition measures immediately after (after recovery intervention) and at 24, 36, 48 hours after the recovery intervention.

ELIGIBILITY:
Inclusion Criteria:

* Elite young professional football players
* 75 minutes (at least) of game participation

Exclusion Criteria:

* Goalkeepers
* Injured players
* Players unable to perform at their best
* Players under medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Neuromuscular or physical performance measures change: jump height | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Counter Movement Jump (CMJ) will be performed to determine the maximum height in centimeters (cm). From standing position with the hands fixed on the hips, participants will be required to bend their knees to a freely chosen angle and perform a maximal vertical jump. Participants will be instructed to keep their body vertical throughout the jump, and to land with knees fully extended. Any jump that will be perceived to deviate from the required instructions will be repeated. Players will jump 3 times as high as possible and the average of the three jumps will be used in subsequent analysis. A 30-s passive recovery phase will be provided between jumps.
Neuromuscular or physical performance measures change: maximal voluntary isometric contraction (MVIC) | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Isometric Hamstring Strength (IHS). Players will be in a supine position, with the tested leg strapped around the ankle (in a neutral position) and performed a hip extension (with a slight knee flexion 20º, while the non-dominant leg was resting on the floor). Players will place their hands on the wall to avoid sliding on the floor. A strain gauge will be placed between the ankle strap and the cord to evaluate the force (MVIC) exerted at a sampling frequency of 80Hz (Chronojump, Boscosystem®️, Barcelona, Spain).
  The tester will give all participants the same instructions; "to exert maximal force down to the floor" and continuous and standardized verbal motivation for 5 seconds. Each limb will be tested 3 times, in a randomized order. The assessment of both legs will be separated by 30 seconds while the time separating two trials of the same leg will be 60 seconds . The MVIC will be tested and measured in Newtons (N).
Biochemical/Physiological measures change: creatine kinase | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Creatine Kinase (CK): units/L
Biochemical/Physiological measures change: mioglobin | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Mioglobin: n/mol/L
Biochemical/Physiological measures change: urea | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Urea: umol/L or mg/dL
Biochemical/Physiological measures change: ions | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Na and K ions: mmol/L

SECONDARY OUTCOMES:
Range Of Movement (ROM) measures change: internal rotation of the hip | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Internal rotation of the hip test will be performed to determine the maximum rotation (º) degrees of this joint. Players will lie down (prone position), with legs stretched out. They will put their leg at 90 degrees and allow that leg to flop out to the side, making sure to keep the opposite hip firmly on the ground. From here, the angle that their leg can rest outward will be assessed. It will be performed and recorded two times for each leg and the average will be used.
Range Of Movement (ROM) measures change: ankle dorsiflexion degrees | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Ankle dorsiflexion test will be performed to determine the maximum range of movement of this joint. This test needs to be done against a wall. Players will be asked to place their foot in a way that an imaginary line drawn through the heel and big toe will be aligned on the tape measure on the floor. Players will be instructed to lunge forward until their knee touches the wall. The heel will be required to remain in contact with the floor at all times. The foot will be moved away from the wall to the point where the knee will only make slight contact with the wall. The leg not being tested will rest on the floor and participants won't be allowed to hold onto the wall for support. The dorsiflexion range of movement will be measured in degrees (º) and the average of two attempts will be used.
Range Of Movement (ROM) measures change: hamstrings extension ASLR | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Active Straight Leg Raise (ASLR) test will be performed to determine the maximum extension (º) degrees of this muscle group. Players will lie down (supine position), with the knees over the mat. Once positioned, the players will be asked to slowly raise their limb with the knee fully extended and the ankle in maximal dorsiflexion. During the test, the non-tested limb will keep on the mat, with the ankle in maximum dorsiflexion and the head on the ground. When the maximum ROM will be reached, the angle that their leg will achieve will be assessed. It will be performed and recorded two times for each leg and the average of two attempts will be used.
Range Of Movement (ROM) measures change: hamstrings extension Jurdan | Baseline, Immediately after intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Jurdan Test will be performed. Initially, the player will be in supine in a similar position to the modified Thomas test but will be asked to complete an active knee extension (holding the thigh at 90°) while holding the table and holding the lumbar spine in contact with the table. The lumbar position will be verified kinaesthetically by the practitioner in the starting position and visually during execution. Maintenance of the thigh angle at around 90° for the active knee extension during testing will be visually verified. The result will be defined as the difference between the actively lengthened legs shin angle and the opposite legs passive thigh angle (which is hanging over the table's edge). Both angles (º degrees) will be measured relative to horizontal. It will be performed and recorded two times for each leg and the average of the two attempts will be used.
Subjective perceptual/well-being questionnaire measures change: McLean | Baseline, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  The questionnaire (McLean et al. 2010) will assess participants' fatigue, sleep quality, general muscle soreness, stress levels and mood on a five-point scale (scores of 1 to 5, 0.5 point increments, being 5 the best state and 0 the worst). Overall well-being will then be determined by summing the five scores.
Subjective perceptual/well-being questionnaire measures change: recovery | Baseline, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Total Quality Recovery Perceived (TQRper) using a 10 point Borg scale (being 0 extremely tired/very poorly recovered and 10 highly energetic/very well recovered) will also be recorded.
Subjective perceptual/well-being questionnaire measures change: RPE | After intervention, 24 hours after intervention, 48 hours after intervention, 72 hours after intervention
  Rate of Perceived Exertion (RPE) using the Foster 0-10 scale (being 0 no exertion and 10 maximal exertion) will also be recorded. Players will respond one simple question: How hard was your session? Each player will complete the 0-to-10 scale without the presence of other players and will not see the values of other participants. Players will be allowed to mark a plus sign (interpreted as 0.5 point) alongside the integer value

CONTACTS AND LOCATIONS:
Overall Officials: Albert Altarriba-Bartes, Principal Investigator — UVic-UCC
Locations (1):
- Universitat de Vic-Universitat Central de Catalunya, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McLean BD, Coutts AJ, Kelly V, McGuigan MR, Cormack SJ. Neuromuscular, endocrine, and perceptual fatigue responses during different length between-match microcycles in professional rugby league players. Int J Sports Physiol Perform. 2010 Sep;5(3):367-83. doi: 10.1123/ijspp.5.3.367. PMID 20861526